CLINICAL TRIAL: NCT01416493
Title: An OPEN LABEL Phase II Safety Study of Bovine Intestinal Alkaline Phosphatase (bIAP), an Inflammation Modulating Moiety, in RA Patients
Brief Title: Bovine Intestinal Alkaline Phosphatase (bIAP) Modulating Rheumatoid Arthritis
Acronym: ALS-003-2008
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alloksys Life Sciences B.V. (Industry)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REUMAP; 2008-007346-63 (EudraCT Number)
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Acute Rheumatoid Arthritis
Keywords: acute rheumatoid arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bIAP treatment (Experimental)
  Interventions: Drug: s.c. injections of bovine intestinal Alkaline Phosphatase

INTERVENTIONS:
Drug: s.c. injections of bovine intestinal Alkaline Phosphatase — daily subcutaneous treatment with two injections of 2000IU bIAP for three days

SUMMARY:
This is a proof of concept study asking if alkaline phosphatase injections can reduce acute inflammation in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This is a proof of concept study to establish the safety of subcutaneous (sc) treatment and the efficacy of alkaline phosphatase (AP) in reducing specific pro-inflammatory cytokines during and after 3 days of twice daily s.c. treatment. A total dose of 12000 Units AP will be administered by 2000 IU s.c. injection twice daily for 3 days. Subjects will be closely followed for 8 days and regular clinical observations will be made during 3 months. Close out will be 3 months after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients of any race with an age >18 years. Woman of child-bearing potential must be on regular contraceptives throughout the trial (Pregnancy tests).

1A: RA according to the 1987 revised ARA criteria (Arnett 1987) with an active disease with DAS28>3.2 despite the prior or concurrent use of DMARDs.

2. Patients may be on no active therapy or may be on continuous DMARD therapy including Methotrexate, Sulphasalazine, Leflunomide, Hydroxychloroquine, Myocrisin alone or in combination, or on NSAID treatment, or on steroid (prednisolone not more than 10mg/day).

3. Patients must have a measurable acute phase response: CRP (> 10mg/dl), ESR > 25. (to be measured on routine lab range CRP/ ESR/AP/ standard biochemistry)

4. Patients eligible for treatment with biological TNFα blockers and who are awaiting the administration of such treatment may enroll in the laboratory and safety protocols Data for Clinical Phase observations will be collected but will be handled as last observation carried forward for the final records prior to the administration of TNF blocking agent, should that occur within the 3-month Clinical Phase. The administration of TNFα blockers will not be delayed for the protocol.

5. Patients who have given written informed consent prior to participation in the trial and who undertake to comply with the protocol.

Exclusion Criteria:

1. Patients who are unwilling or unable to be fully evaluated for follow-up.
2. Patients who have an active infection or who are suspected of having systemic infection and or patients that are treated with antibiotics.
3. Patients whose screening blood do not reflect a sufficient cytokine or acute phase response.
4. Patients who have evidence of significant hepatic disease, including history of clinical signs or laboratory values of total bilirubin > 34.2 umol/L (> 2.0 mg/dL), ALT (>120) or AST (>135) corresponding to > 3X upper limit of normal.
5. Alkaline phosphatase levels must be less 145 IU/L (routine clinical method)
6. Patients who received investigational drugs in the 30 days prior to study drug administration, or are currently participating in a study during which the administration of investigational drugs within one month is anticipated.
7. Patients who have renal insufficiency (history of creatinine >177umol/L or >2.0 mg/dL) or chronic renal failure requiring dialysis.
8. Patients with severe neurological deficits (see Appendix I).
9. Patients who have a recent history of drug substance or alcohol abuse.
10. Patients with a diagnosis of idiopathic thrombocytopenia.
11. Patients with a history of cancer who have received chemotherapy or radiation therapy within the past 3 months. Patients receiving only adjuvant hormonal therapy are not excluded. If the cancer has not resolved completely, the patient should not be enrolled without permission of Alloksys.
12. Patients receiving oral glucocorticoids >10mg /day or any IV, IM or Intra articular dosing within 30 days of commencing the protocol.
13. Patients who are vegetarians or veganists or those patients that may be expected not to be tolerant to bovine proteins, or not to wish exposure to bovine proteins for personal reasons.
14. Patients who are, in the opinion of the Investigator or the Sponsor, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
blood level of the pro-inflammatory cytokines: TNFα and IL6 | 3 months
  The anticipated effects of bIAP will be short lived, within 4 days. However, in order to capture durable clinical responses or any late adverse effects, patients will be followed through 3 months at weeks 2, 4, 8 and 12 incorporating trial observations with routine monthly care to reduce disruption to patients.

SECONDARY OUTCOMES:
RA clinical status expressed as Daily Activity Score (DAS-28) | 3 months
  van der Heijde DM, van 't Hof MA, van Riel PL, Theunisse LA, Lubberts EW, van Leeuwen MA, van Rijswijk MH, van de Putte LB. Judging disease activity in clinical practice in rheumatoid arthritis: first step in the development of a disease activity score. Ann Rheum Dis. 1990 Nov;49(11):916-920

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hammond, MD, Principal Investigator — Maidstone Hospital, Dept. Rheumatology
Locations (1):
- Maidstone Hospital, Dept. Rheumatology, Maidstone, Kent, United Kingdom

REFERENCES:
- See also: an other running study with bovine Intestinal Alkaline Phosphatase (bIAP) — http://clinicaltrials.gov/ct2/show/NCT01144611